CLINICAL TRIAL: NCT01052363
Title: OXC401-PO1s/WVU 1309 - A Pilot Study of Fosbretabulin With Bevacizumab in Recurrent High-Grade Gliomas
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No funding
Sponsor: West Virginia University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WVU1309
Record Dates: First submitted 2010-01-19; First posted 2010-01-20 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Central Nervous System Tumors
Keywords: CNS tumors
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CA4P + Avastin (Experimental)
  Interventions: Drug: Bevacizumab, CA4P
- Avastin + CA4P (Experimental)
  Interventions: Drug: Bevacizumab, CA4P

INTERVENTIONS:
Drug: Bevacizumab, CA4P

SUMMARY:
Pilot Trial of CA4P with Avastin in Recurrent Gliomas

DETAILED DESCRIPTION:
The purpose of this study is to see if fosbretabulin, the drug being studied, combined with bevacizumab will help your brain cancer and if using these drugs together is safe.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed grade III Anaplastic gliomas (including anaplastic astrocytoma, anaplastic oligodendroglioma, and anaplastic oligoastrocytoma) or Grade IV Glioblastoma multiforme.
2. Recurrence or progression after failing first line treatment of temozolomide chemotherapy and radiation. Patient who failed additional lines of treatment are eligible for participating in the trial. Patients must have measurable disease, defined as having contrast enhancing measurable disease on MRI of brain. Baseline MRI should be done no more than 2 weeks from starting treatment.
3. At least 4 weeks since prior chemotherapy or radiation therapy, 4 weeks if the last regimen included BCNU.
4. Age greater than 18 years. Because no dosing or adverse event data are currently available on the use of fosbretabulin in combination with bevacizumab in patients less than 18 years of age, children are excluded from this study.
5. Life expectancy of greater than 3 months.
6. ECOG performance status 0-2 Karnofsky greater than 60%).
7. Patients must have normal organ and marrow function as defined.
8. The effects of fosbretabulin on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because vascular disrupting agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant (including female partners of male study participants) or suspect she is pregnant while participating in this study, she should inform the Investigator and her treating physician immediately.
9. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
2. Patients with prior treatment using bevacizumab.
3. Patients should not have received any other investigational agents within 4 weeks.
4. History of abdominal fistula, GI perforation or intra-abdominal abscess within the last 6 months.
5. Coagulopathy or bleeding diathesis. Patients on therapeutic dose of anticoagulation are excluded from the study.
6. Uncontrolled intercurrent illness including, but not limited to, ongoing active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. Also, MI/unstable angina within 6 months; stroke/TIA within 1 year; symptomatic claudication within 1 year; abnormalities on ECG including prolonged QTc interval (i.e. > 450 ms for males and > 470 ms for females), new Q-wave, RBBB, LBBB,ST-segment depression.
7. Grade 3 proteinuria (> 3.5 g protein/24 hours)
8. Uncontrolled hypertension (blood pressure >150/100 during Screening)
9. Clinically significant peripheral vascular disease.
10. History of allergic reactions attributed to compounds of similar chemical or biologic composition to fosbretabulin or other agents used in the study.
11. Since dilantin induces the P450 system and the effect this will have on fosbretabulin or bezvacazimab is not known, patients that are on seizure prophylaxis with dilantin will not be eligible. Switching the seizure prophylaxis to noninducers of the P450 system such as levetiracetam is acceptable. Patients must be off dilantin for one week before starting this clinical trial. Additionally fosbretabulin has the potential to interact with drugs metabolized by CYP2C19 which includes barbiturates, diazepam and valproic acid. However the clinical significance of these interactions is not known.
12. Pregnant women are excluded from this study because fosbretabulin is a vascular disrupting agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with fosbretabulin, breastfeeding should be discontinued if the mother is treated with fosbretabulin.
13. HIV-positive patients on combination antiretroviral therapy are ineligible Because of the potential for pharmacokinetic interactions with fosbretabulin. In addition,these patients are at increased risk of lethal infections when treated with marrowsuppressive therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01

CONTACTS AND LOCATIONS:
Overall Officials: Ramin Altaha, MD, Principal Investigator — West Virginia University
Locations (1):
- MBRCC, West Virginia University, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No